CLINICAL TRIAL: NCT00002504
Title: OUTPATIENT SUBCUTANEOUS IL-2 AND ALPHA INTERFERON IN THE MANAGEMENT OF METASTATIC CANCER
Brief Title: Interleukin-2 Plus Interferon Alfa in Treating Adults With Metastatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Collaborators: Cancer Biotherapy Research Group (Other)
Responsible Party: Robert O. Dillman, MD, Hoag Memorial Hospital Presbyterian
Purpose: Treatment
Other Study IDs: CDR0000077942; CBRG-9211; NBSG-9211; NCI-V92-0148
Record Dates: First submitted 1999-11-01; First posted 2004-07-26 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous/Nonmalignant Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; monoclonal gammopathy of undetermined significance; recurrent adult Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; polycythemia vera; chronic idiopathic myelofibrosis; essential thrombocythemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; prolymphocytic leukemia; primary systemic amyloidosis; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Hodgkin Disease; Monoclonal Gammopathy of Undetermined Significance; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone | interventions — aldesleukin; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alfa

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill metastatic cancer cells. Interferon alfa may interfere with the growth of the cancer cells. Combining interleukin-2 and interferon alfa may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of interleukin-2 plus interferon alfa in treating adults with metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, failure-free survival, and overall survival of interleukin-2 and interferon alpha administered subcutaneously on an outpatient basis for 8 weeks to patients with metastatic cancer. II. Determine the toxicities associated with this therapy.

OUTLINE: Biological Response Modifier Therapy. Interleukin-2 (Cetus), IL-2, NSC-373364; Interferon alpha (Schering), IFN-A, NSC-377523.

PROJECTED ACCRUAL: Up to 30 patients with various malignancies will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic cancer of any type Measurable or evaluable disease required, i.e.: Bidimensionally measurable lesions on physical exam, x-ray, CT, MRI, or other radiologic procedure Any lesion apparent on radiologic exam that is not measurable in 2 perpendicular diameters Previously irradiated lesions acceptable provided subsequent progression is documented No active brain metastases Previously treated brain metastases allowed provided measurable/evaluable disease exists outside the CNS

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Hematopoietic: (within 14 days prior to entry) WBC at least 3,000 Platelets at least 100,000 Hematocrit at least 30% (may be transfused) Hepatic: (within 14 days prior to entry) Bilirubin less than 2.0 mg/dl PT and PTT normal Renal: (within 14 days prior to entry) Creatinine less than 2.0 mg/dl Cardiovascular: No MI within 6 months No medication for arrhythmia No medication for CHF Hypertension that is stable off medication allowed Pulmonary: pO2 at least 60 mm Hg in patients with primary lung cancer or symptomatic pulmonary disease Reasonable respiratory reserve No dyspnea at rest No requirement for supplemental oxygen Other: No familial history of malignant hyperthermia No chronic underlying immunodeficiency disease No HIV seropositivity No active infection requiring antibiotic therapy No other serious intercurrent illness No concurrent malignancy No pregnant or nursing women Adequate contraception required of fertile women

PRIOR CONCURRENT THERAPY: No concurrent therapy with other anticancer agents No concurrent immunosuppressive agents (e.g., cyclosporin) Biologic therapy: Prior interferon alpha allowed Chemotherapy: At least 4 weeks since systemic chemotherapy with recovery required Endocrine therapy: No concurrent corticosteroids Radiotherapy: At least 4 weeks since radiotherapy Surgery: Adequate recovery required Other: No prior organ allograft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1992-08; Primary Completion 1998-02 (Actual); Study Completion 1999-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Cancer Biotherapy Research Group
Locations (5):
- United States (5):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Bloomington Hospital, Bloomington, Indiana
  - St. Vincent Hospital and Health Care Center Research Department, Indianapolis, Indiana
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee

REFERENCES:
- [Result] Dillman RO, Soori G, Tai DF, et al.: Outpatient subcutaneous (SC) interleukin-2 (IL-2) and interferon alpha (IFN) in the management of metastatic cancer: a preliminary report. J Immunother 20(5): 404, 1997.